CLINICAL TRIAL: NCT00230399
Title: C-2424: Phase II Study of Celecoxib, Capecitabine, and Irinotecan in Patients With Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy Treatments in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Dr. Mark Zalupski, University of Michigan Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 3-24
Record Dates: First submitted 2005-09-09; First posted 2005-09-30 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib; Capecitabine; Irinotecan

INTERVENTIONS:
Drug: Celecoxib
Drug: Capecitabine
Drug: Irinotecan

SUMMARY:
This study will examine a new combination of drugs: celecoxib, capecitabine and irinotecan, for the treatment of metastatic colorectal cancer. Capecitabine and irinotecan, individually, are approved by the Food and Drug Administration (FDA) for use in colorectal cancer. The combination of these two drugs is experimental (not approved by the FDA as standard treatment), but is a widely used treatment option and preliminary studies have shown that treatment with the combination of capecitabine and irinotecan has a positive effect on metastatic colorectal cancer. Likewise, previous research in animals has shown that celecoxib, a drug approved for arthritis therapy, also has activity against this tumor type and may improve the anti-cancer activity of the combination of capecitabine and irinotecan.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a histologically proven adenocarcinoma of colon or rectum with metastases or local recurrence.
2. Patients must have at least one measurable lesion according to the RECIST criteria. Bone metastases, ascites and pleural effusion are not measurable.
3. Minimum indicator lesion size as follows:

   Greater than or equal to 20 mm measured by conventional CT Greater than or equal to 10 mm measured by spiral techniques
4. Prior use of celecoxib for the treatment of nonmalignant disorders is allowed.
5. Patients must have a performance status of 0,1, or 2 by the Southwest Oncology Group criteria.
6. Patients must have a calculated creatinine clearance of greater than 50 ml/min.
7. Patients must have an absolute neutrophil count of greater than or equal to 1500/ml, platelet count greater than or equal to 100,000/ml, and total serum bilirubin equal or less than the institution's upper limit or normal range.
8. Patients must have recovered from any effects of surgery.
9. Evaluable disease must be present outside radiation field. At least 3 weeks must have elapsed after discontinuation of radiation therapy.
10. Patients must provide a signed consent to participate in the study.

Exclusion Criteria:

1. Patients with a proven history of peptic ulcer disease or gastroesophageal reflux.
2. Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other non-steroidal anti-inflammatory drugs.
3. Patients who have received prior chemotherapy for colorectal cancer (including capecitabine or irinotecan) except for patients relapsing more than 6 months after completion of adjuvant chemotherapy.
4. History of other malignancy, except for cancers that have been treated with a curative intent and patient is without evidence of active disease.
5. Unresolved bacterial infection requiring treatment with antibiotics.
6. Pregnant or lactating women may not participate in the study. Women/men of reproductive age group may not participate unless they have agreed to use an effective method of contraception.
7. Patients who have allergy to any of the study drugs or sulfa drugs.
8. Patients known to have HIV-1 virus infection because of the undetermined effect of this chemotherapy regimen in patients with HIV-1 and the potential for serious interaction with anti-HIV medications.
9. Gilbert's disease.
10. Lack of physical integrity of the upper gastrointestinal tract. Inability to swallow tablets or those who have malabsorption syndrome.
11. Other serious concurrent infection
12. Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-06; Primary Completion 2006-01 (Actual); Study Completion 2008-03

PRIMARY OUTCOMES:
To determine the objective response rate to the combination of celecoxib, capecitabine, and irinotecan in patients with metastatic colorectal cancer.

SECONDARY OUTCOMES:
To evaluate the time to progression of metastatic colorectal cancer after treatment with celecoxib, capecitabine, and irinotecan.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States